CLINICAL TRIAL: NCT05417620
Title: Optimizing Pre-exposure Prophylaxis (PrEP) Implementation and Effectiveness Among Women at High Risk for HIV Acquisition in South Africa
Brief Title: Le Kip Kip: A Campaign to Change Social Norms and Build Sustainable Demand for PrEP Among Women in South Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); TB HIV Care (Other); Community Media Trust (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 90089975; R01MH121161 (NIH)
Record Dates: First submitted 2022-06-02; First posted 2022-06-14 (Actual); Results first posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Pre-exposure Prophylaxis; HIV Infections
Keywords: PrEP; Pre-exposure Prophylaxis; HIV prevention; Cluster randomized trial; Community-based methods; Key populations; Female sex workers; Adolescent girls and young women; South Africa
MeSH Terms: conditions — HIV Infections | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Standard of Care (Other): Full-time peer educators employed by the TB HIV Care programme to engage women, layer PrEP promotion across prevention programs, and implement "refer a friend" strategies, information, education and communication (IEC) materials, service user testimonials, risk reduction posters to increase young women's perception of risk, working after hours/weekends to reach young women, working with school governing bodies, and door-to-door outreach.
  Interventions: Other: Standard of Care
- Enhanced social media campaign (Experimental): Social media campaign which will be disseminated on Facebook, Instagram, and WhatsApp with targeted ads/promotion of materials in intervention districts.
  Interventions: Behavioral: Social Media Campaign
- Enhanced social media campaign + PrEP champions (Experimental): Venue-based peers who will provide PrEP information, share personal experiences with PrEP, and refer young women to TB HIV Care to receive PrEP if interested in addition to the enhanced social media campaign.
  Interventions: Behavioral: Social Media Campaign; Behavioral: PrEP Champions
- Enhanced social media campaign + Community mobilization (Experimental): Peers will work within wards to organize and attend community meetings to share PrEP information and facilitate discussions with young women, male partners, family members, and other community members in addition to the enhanced social media campaign.
  Interventions: Behavioral: Social Media Campaign; Behavioral: Community Mobilization
- Enhanced social media campaign + PrEP champions + Community mobilization (Experimental): Clusters in this arm will receive both the PrEP champion and community mobilization interventions in addition to the enhanced social media campaign.
  Interventions: Behavioral: Social Media Campaign; Behavioral: PrEP Champions; Behavioral: Community Mobilization

INTERVENTIONS:
Behavioral: Social Media Campaign — PrEP social influence campaign, which will use online approaches to promote PrEP within communities in addition to the standard of care activities. Messaging crafted with community input will be geographically targeted to women, parents/mentors, and male partners on Facebook, Instagram, and Whatsapp, all with the intention to promote PrEP for women at high risk of HIV infection and change community norms and influence around PrEP. A combination of static imagery and brief videos will be used to engage these groups via social media platforms. A Facebook page will be created and maintained that can be accessed by anyone anywhere, but will only be advertised/promoted in the intervention districts.
  Arms: Enhanced social media campaign; Enhanced social media campaign + Community mobilization; Enhanced social media campaign + PrEP champions; Enhanced social media campaign + PrEP champions + Community mobilization
Behavioral: PrEP Champions — Within venues served by the FSW and AGYW programs, the team will identify and train 1 venue-based PrEP champion per venue who will receive supplies (e.g. a hat, pin and posters, flyers, IEC material) to wear to promote PrEP, facilitate linkage between women interested in PrEP and the TB HIV Care PrEP programme. PrEP champions will be either peers with experience taking PrEP, venue managers or local influencers (e.g. women running shops next to the mobile serving AGYW) that have repeated contact with the women the programme is intended to serve. The final selection of PrEP champions will be made in consultation with the Community Advisory Groups, venues and by the programme who works closely with each of the sites.
  Arms: Enhanced social media campaign + PrEP champions; Enhanced social media campaign + PrEP champions + Community mobilization
Behavioral: Community Mobilization — A PrEP community mobilization team (2 peers, including one woman and one man) will be recruited within each ward to promote PrEP. The team will present information about PrEP and the PrEP programme at the ward councilors meeting, at Learning Support Agent meetings with parents/guardians, at local events/fairs, community meetings and through engaging men, women and parents across the community through informal conversations. Teams will be wearing branded material and will focus on presenting factual information and decreasing PrEP stigma. Each team will focus on promoting PrEP within their own ward over the 6-month period.
  Arms: Enhanced social media campaign + Community mobilization; Enhanced social media campaign + PrEP champions + Community mobilization
Other: Standard of Care — Full-time peer educators employed by the TB HIV Care programme to engage women, layer PrEP promotion across prevention programs, and implement "refer a friend" strategies, information, education and communication (IEC) materials, service user testimonials, risk reduction posters to increase young women's perception of risk, working after hours/weekends to reach young women, working with school governing bodies, and door-to-door outreach.
  Arms: Standard of Care

SUMMARY:
The purpose of this study is to evaluate the impact of a social media campaign and community engagement activities to promote pre-exposure prophylaxis (PrEP) use among young women and to influence community norms around PrEP in South Africa. To do this, the investigative team will analyze PrEP initiation and retention data from the study's implementing partner, TB HIV Care, a non-profit organization providing PrEP to marginalized young women in South Africa. The effect of the social media campaign and community engagement will be tested using a short duration cluster randomized trial (CRT).

DETAILED DESCRIPTION:
The cluster randomized trial (CRT) will not engage in PrEP provision to individuals, but instead employs geographical regions to serve as units of randomization where social media content and community engagement will be targeted. TB HIV Care employs a large team to provide routine service delivery while the CRT tests strategies including a social media campaign and community engagement that may amplify PrEP uptake and persistence among the community, leveraging the programme infrastructure to actually provide services as it is already doing. Embedding strategies within the programme ensures that the existing results come from real world contexts and focuses on implementation of support strategies rather than clinical care provision. The CRT will be implemented across 10 districts, with 5 districts serving as control sites and 5 as intervention sites.

ELIGIBILITY:
Inclusion Criteria:

* Eligible to take PrEP per TB HIV Care programmatic criteria
* Engaged in TB HIV Care HIV prevention program

Exclusion Criteria:

* Not eligible for PrEP (not at risk for HIV) per TB HIV Care programmatic criteria

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Eligibility to limited to cisgender women
Enrollment: 601 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheree R Schwartz, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- TB HIV Care, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: No
Aggregate programmatic data will be used to assess trial outcomes rather than individual participant data given the cluster randomized trial design. Therefore, no individual participant data (IPD) will be collected and no sharing plan is required.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 601 participants were enrolled and engaged in HIV prevention services from the TB HIV Care Program. The TB HIV Care program had a total of 25,168 service-users in their database who initiated prep and were included in the analysis.
Units Other Than Participants: wards
Groups:
- Enhanced Social Media Campaign: Social Media Campaign: PrEP social influence campaign, which will use online approaches to promote PrEP within communities in addition to the standard of care activities. A combination of static imagery and brief videos will be used to engage these groups via social media platforms. A Facebook page will be created and maintained that can be accessed by anyone anywhere, but will only be advertised/promoted in the intervention districts.
- Enhanced Social Media Campaign + PrEP Champions: Social Media Campaign: PrEP social influence campaign, which will use online approaches to promote PrEP within communities in addition to the standard of care activities. A combination of static imagery and brief videos will be used to engage these groups via social media platforms. A Facebook page will be created and maintained that can be accessed by anyone anywhere, but will only be advertised/promoted in the intervention districts.
  PrEP Champions: Venue-based PrEP champions will receive supplies (e.g. a hat, pin and posters, flyers, IEC material) to wear to promote PrEP, facilitate linkage between women interested in PrEP and the TB HIV Care PrEP programme. PrEP champions will be either peers with experience taking PrEP, venue managers or local influencers that have repeated contact with the women the programme is intended to serve.
- Enhanced Social Media Campaign + Community Mobilization: Social Media Campaign: PrEP social influence campaign, which will use online approaches to promote PrEP within communities in addition to the standard of care activities. A combination of static imagery and brief videos will be used to engage these groups via social media platforms. A Facebook page will be created and maintained that can be accessed by anyone anywhere, but will only be advertised/promoted in the intervention districts.
  Community Mobilization: PrEP community mobilization teams will be recruited to promote PrEP. The team will present information about PrEP and the PrEP programme at the ward councilors meeting, Learning Support Agent meetings with parents/guardians, local events/fairs, community meetings and through engaging men, women and parents across the community through informal conversations. Teams will be wearing branded material and will focus on presenting factual information and decreasing PrEP stigma.
- Enhanced Social Media Campaign + PrEP Champions + Community Mobilization: Social Media Campaign: PrEP social influence campaign, which will use online approaches to promote PrEP within communities in addition to the standard of care activities. A combination of static imagery and brief videos will be used to engage these groups via social media platforms. A Facebook page will be created and maintained that can be accessed by anyone anywhere, but will only be advertised/promoted in the intervention districts.
  PrEP Champions: Venue-based PrEP champions will receive supplies (e.g. a hat, pin and posters, flyers, IEC material) to wear to promote PrEP, facilitate linkage between women interested in PrEP and the TB HIV Care PrEP programme. PrEP champions will be either peers with experience taking PrEP, venue managers or local influencers that have repeated contact with the women the programme is intended to serve.
  Community Mobilization: PrEP community mobilization teams will be recruited to promote PrEP. The team will present information about PrEP and the PrEP programme at the ward councilors meeting, Learning Support Agent meetings with parents/guardians, local events/fairs, community meetings and through engaging men, women and parents across the community through informal conversations. Teams will be wearing branded material and will focus on presenting factual information and decreasing PrEP stigma.
Period: Overall Study
Arm/Group | Standard of Care | Enhanced Social Media Campaign | Enhanced Social Media Campaign + PrEP Champions | Enhanced Social Media Campaign + Community Mobilization | Enhanced Social Media Campaign + PrEP Champions + Community Mobilization
Started | 301; 50 wards | 92; 27 wards | 55; 26 wards | 48; 26 wards | 105; 26 wards
Service-users in the TB HIV Care Program Database at the Ward-level (Not Enrolled) | 17949; 50 wards | 3091; 27 wards | 924; 26 wards | 925; 26 wards | 2279; 26 wards
Completed | 301; 50 wards | 92; 27 wards | 55; 26 wards | 48; 26 wards | 105; 26 wards
Not Completed | 0; 0 wards | 0; 0 wards | 0; 0 wards | 0; 0 wards | 0; 0 wards

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were analyzed for 601 service-users surveyed pre-intervention from three selected control districts (n=301) and randomized wards within three selected intervention districts (n=300) to assess service-user characteristics before the intervention.
Units Other Than Participants: Wards
Groups:
- Enhanced Social Media Campaign/PrEP Champions/Community Mobilization: PrEP social influence campaign, which will use online approaches to promote PrEP within communities in addition to the standard of care activities. A combination of static imagery and brief videos will be used to engage these groups via social media platforms. A Facebook page will be created and maintained that can be accessed by anyone anywhere, but will only be advertised/promoted in the intervention districts.
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Enhanced Social Media Campaign/PrEP Champions/Community Mobilization | Enhanced Social Media Campaign + PrEP Champions | Enhanced Social Media Campaign + Community Mobilization | Enhanced Social Media Campaign + PrEP Champions + Community Mobilization | Total
Number analyzed (Participants) | 301 | 92 | 55 | 48 | 105 | 601
Number analyzed (Wards) | 50 | 27 | 26 | 26 | 26 | 155
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.8 (7.8) | 26.4 (7.8) | 28.2 (8.8) | 25.2 (7.8) | 24.7 (7.2) | 24.9 (7.9)
Age, Customized [Count of Participants; unit: Participants]
  Age: 15-17 | 80 | 9 | 2 | 7 | 12 | 110
  Age: 18-24 | 117 | 37 | 21 | 18 | 51 | 244
  Age: 25-29 | 33 | 17 | 7 | 14 | 20 | 91
  Age: 30-34 | 32 | 13 | 11 | 4 | 12 | 72
  Age: 35+ | 39 | 16 | 14 | 5 | 10 | 84
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 301 | 92 | 55 | 48 | 105 | 601
  Male | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 297 | 92 | 54 | 47 | 104 | 594
  White | 3 | 0 | 0 | 0 | 0 | 3
  More than one race | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Africa | 301 | 92 | 55 | 48 | 105 | 601
Education Level [Count of Participants; unit: Participants] — Population: Row population differs from the overall as participants had the option to skip or decline to answer certain questions.
  Participants
    number analyzed (Participants) | 293 | 82 | 45 | 47 | 102 | 569
    Currently in school | 142 | 26 | 15 | 11 | 57 | 251
    Did not complete highschool | 36 | 16 | 9 | 10 | 17 | 88
    Completed highschool | 93 | 31 | 17 | 21 | 24 | 186
    Completed university/trade school or higher | 22 | 9 | 4 | 5 | 4 | 44
Relationship Status [Count of Participants; unit: Participants] — Population: Row population differs from the overall as participants had the option to skip or decline to answer certain questions.
  Participants
    number analyzed (Participants) | 300 | 92 | 54 | 45 | 105 | 596
    Single | 126 | 32 | 23 | 13 | 32 | 226
    Steady partner not living together | 169 | 39 | 14 | 20 | 58 | 300
    Steady partner living together | 5 | 21 | 17 | 12 | 15 | 70
Current Housing Status [Count of Participants; unit: Participants] — Population: Row population differs from the overall as participants had the option to skip or decline to answer certain questions.
  Participants
    number analyzed (Participants) | 297 | 91 | 55 | 48 | 104 | 595
    Owns/rents | 66 | 30 | 23 | 14 | 32 | 165
    Staying with others (e.g., family, friends) | 200 | 56 | 29 | 34 | 59 | 378
    Shelter | 9 | 0 | 0 | 0 | 1 | 10
    Student housing | 5 | 5 | 3 | 0 | 12 | 25
    Brothel | 17 | 0 | 0 | 0 | 0 | 17
Currently Taking PrEP [Count of Participants; unit: Participants] — Population: Row population differs from the overall as participants had the option to skip or decline to answer certain questions.
  Participants
    number analyzed (Participants) | 301 | 92 | 55 | 48 | 104 | 600
    (all) | 133 | 58 | 43 | 27 | 59 | 320
Smartphone Ownership [Count of Participants; unit: Participants] | 224 | 66 | 40 | 29 | 74 | 433
Participants With Internet Access [Count of Participants; unit: Participants] — Population: Row population differs from the overall as participants had the option to skip or decline to answer certain questions.
  Participants
    number analyzed (Participants) | 300 | 89 | 55 | 48 | 104 | 596
    (all) | 218 | 69 | 36 | 30 | 78 | 431

OUTCOME MEASURES:

1. Primary Outcome: Number of Service-users Who Initiate PrEP Uptake Within the TB HIV Care Programme
Description: De-identified aggregate counts of female sex workers (FSW) and adolescent girls and young women (AGYW) service-users within the TB HIV Care programme database who initiate PrEP during the intervention period. Number of service users in the program database who initiated prep are reported.
Time Frame: 12 months
Population: The analysis population are de-identified aggregate FSW and AGYW service-users in the TB HIV Care program database that initiated PrEP during the study period.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Enhanced Social Media Campaign | Enhanced Social Media Campaign + PrEP Champions | Enhanced Social Media Campaign + Community Mobilization | Enhanced Social Media Campaign + PrEP Champions + Community Mobilization
Number analyzed (Participants) | 17949 | 3091 | 924 | 925 | 2279
Participants | 17949 | 3091 | 924 | 925 | 2279
Statistical Analysis 1: Comparison: Standard of Care; This statistical analysis is done at the district level where counts of initiations in intervention districts are compared to standard of care districts. In the measure type we report "rate = average counts of PrEP initiations per number of study months"; Test type: Other; p = 0.707, Regression, Poisson — Threshold for significance: 0.05; Incidence rate ratio = 1.21, 95% CI 2-sided [0.44 to 3.31]

2. Secondary Outcome: Proportion of PrEP Persistence at 1-month Within the TB HIV Care Programme
Description: Proportion of FSW/AGYW clients within the TB HIV Care programme database who return for 1-month follow-up visit. For each district, the proportion of clients who returned for this visit was calculated. The mean proportion across the standard of care and intervention districts is reported.
Time Frame: Month 1
Population: The analysis population are de-identified aggregate FSW and AGYW service-users in the TB HIV Care programme database who initiated PrEP during the trial period and due for a 1-month follow-up visit. The intervention arms are grouped under the social influence campaign intervention as per the study protocol's analytic approach.
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Units Other Than Participants: Districts
Groups:
- Enhanced Social Media Campaign/PrEP Champions/Community Mobilization: Clusters in this arm will receive the enhanced social media campaign alone or combined with PrEP champions, community mobilization, or both.
  Social Media Campaign: PrEP social influence campaign, which will use online approaches to promote PrEP within communities in addition to the standard of care activities. A combination of static imagery and brief videos will be used to engage these groups via social media platforms. A Facebook page will be created and maintained that can be accessed by anyone anywhere, but will only be advertised/promoted in the intervention districts.
  PrEP Champions: Venue-based PrEP champions will receive supplies (e.g. a hat, pin and posters, flyers, IEC material) to wear to promote PrEP, facilitate linkage between women interested in PrEP and the TB HIV Care PrEP programme. PrEP champions will be either peers with experience taking PrEP, venue managers or local influencers that have repeated contact with the women the programme is intended to serve.
  Community Mobilization: PrEP community mobilization teams will be recruited to promote PrEP. The team will present information about PrEP and the PrEP programme at the ward councilors meeting, Learning Support Agent meetings with parents/guardians, local events/fairs, community meetings and through engaging men, women and parents across the community through informal conversations. Teams will be wearing branded material and will focus on presenting factual information and decreasing PrEP stigma.
Arm/Group | Standard of Care | Enhanced Social Media Campaign/PrEP Champions/Community Mobilization
Number analyzed (Participants) | 16769 | 6933
Number analyzed (Districts) | 5 | 5
percentage of participants | 42.88 [8.88 to 76.88] | 27.60 [-9.92 to 65.12]

3. Secondary Outcome: Proportion of PrEP Persistence at 4 Months Within the TB HIV Care Programme
Description: Proportion of FSW/AGYW clients within the TB HIV Care programme database who return for 4-month follow-up visit. For each district, the proportion of clients who returned for this visit was calculated. The mean proportion across the standard of care and intervention districts is reported.
Time Frame: Month 4
Population: The analysis population are de-identified aggregate FSW and AGYW service users in the TB HIV Care programme database who initiated PrEP during the trial period and due for a 4-month follow-up visit. The intervention arms are grouped under the social influence campaign intervention as per the study protocol's analytic approach.
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Units Other Than Participants: Districts
Arm/Group | Standard of Care | Enhanced Social Media Campaign/PrEP Champions/Community Mobilization
Number analyzed (Participants) | 9948 | 4461
Number analyzed (Districts) | 5 | 5
percentage of participants | 29.48 [7.14 to 57.85] | 15.56 [-3.50 to 34.47]

4. Secondary Outcome: Number of Participants Who Found Intervention Acceptable
Description: Acceptability: Respondents who reported intervention acceptability captured in post-trial cross-sectional survey
Time Frame: Month 12
Population: As outlined in the protocol, acceptability of the social media campaign was assessed among post-intervention cross-sectional survey respondents who reported exposure to the Le Kip Kip social influence campaign.
Measure: Count of Participants; unit: Participants
Groups:
- Post-trial Cross-sectional Survey Respondents: FSW and AGYW service users who were enrolled to complete a post-trial cross-sectional survey from selected standard of care and intervention districts.
Arm/Group | Post-trial Cross-sectional Survey Respondents
Number analyzed (Participants) | 153
Participants | 137

5. Secondary Outcome: Adoption as Assessed by Number of Facebook Page Visits by Unique Users
Description: Service user uptake and engagement with campaign measured via the number of Facebook page visits. Facebook users who visited the campaign content is reported.
Time Frame: Month 12
Population: The analysis population is the number Facebook users that have seen the content.
Measure: Number; unit: visits
Groups:
- Le Kip Kip Social Media Campaign: This group consists of individuals who were exposed to the Le Kip Kip Facebook page through organic and paid posts, videos, and page visits.
Arm/Group | Le Kip Kip Social Media Campaign
Number analyzed (Participants) | 631493
visits | 52608

6. Secondary Outcome: Total Cost
Description: Total cost associated with planning, designing, and implementing the social influence campaign will be assessed via review of detailed study budgets. The reported value represents a single point estimate (in USD) of the total cost incurred, based on actual budget expenditures. Because this is a cumulative total cost, non-sampled financial figure, measures of dispersion/precision are not applicable. This outcome measure is based on a review of detailed study budgets related to the planning, design, and implementation of the social influence campaign.The unit analyzed is the campaign itself and analyzed as the overall cost of the Enhanced social media campaign/PrEP champions/Community mobilization arm per protocol.
Time Frame: Month 12
Population: This analysis does not involve any participants
Measure: Number; unit: Dollars
Units Other Than Participants: Social Influence Campaign
Groups:
- Enhanced Social Media Campaign/PrEP Champions/Community Mobilization: Clusters in this arm will receive combinations of the enhanced social media campaign, PrEP champions, and community mobilization.
  Social Media Campaign: PrEP social influence campaign, which will use online approaches to promote PrEP within communities in addition to the standard of care activities. A combination of static imagery and brief videos will be used to engage these groups via social media platforms. A Facebook page will be created and maintained that can be accessed by anyone anywhere, but will only be advertised/promoted in the intervention districts.
  PrEP Champions: Venue-based PrEP champions will receive supplies (e.g. a hat, pin and posters, flyers, IEC material) to wear to promote PrEP, facilitate linkage between women interested in PrEP and the TB HIV Care PrEP programme. PrEP champions will be either peers with experience taking PrEP, venue managers or local influencers that have repeated contact with the women the programme is intended to serve.
  Community Mobilization: PrEP community mobilization teams will be recruited to promote PrEP. The team will present information about PrEP and the PrEP programme at the ward councilors meeting, Learning Support Agent meetings with parents/guardians, local events/fairs, community meetings and through engaging men, women and parents across the community through informal conversations. Teams will be wearing branded material and will focus on presenting factual information and decreasing PrEP stigma.
Arm/Group | Standard of Care | Enhanced Social Media Campaign/PrEP Champions/Community Mobilization
Number analyzed (Participants) | NA | NA
Number analyzed (Social Influence Campaign) | 0 | 1
Dollars |  | 223736

7. Secondary Outcome: Penetration as Assessed by Number of Participants Who Report Engagement With Campaign Among Social Support Networks
Description: Extent to which the social influence campaign reached FSW/AGYW and their families/peers/partners measured via descriptive statistics from post-trial survey questions on campaign exposure and perceptions of the campaign among FSW/AGYW and their social support networks.
Time Frame: Month 12
Population: As outlined in the protocol, penetration of the social influence campaign is captured by post-intervention cross-sectional survey respondents from selected standard of care and intervention districts who answered questions regarding the reach of the Le Kip Kip campaign to their families, peers, and partners.
Measure: Count of Participants; unit: Participants
Arm/Group | Post-trial Cross-sectional Survey Respondents
Number analyzed (Participants) | 600
Participants
  Families: number analyzed (Participants) | 577
  Families | 68
  Peers: number analyzed (Participants) | 576
  Peers | 106
  Partners: number analyzed (Participants) | 560
  Partners | 41

8. Secondary Outcome: Fidelity as Assessed by Percentage of On-Schedule Posts
Description: Extent to which the social influence campaign was carried out according to plan measured via social media metrics to determine whether static and video content were shared across platforms as planned. Fidelity is assessed by tracking adherence to the planned posting schedule. Participants were not included in assessing fidelity of on-schedule posts, rather posts made across social media platforms were analyzed. Adherence was assessed by documenting whether all scheduled posts were successfully and timely published as planned during the campaign period.
Time Frame: Month 12
Population: As outlined in the protocol, participants were not included in assessing fidelity of on-schedule posts, rather posts made across social media platforms were analyzed.
Measure: Count of Units; unit: Posts
Units Other Than Participants: Posts
Groups:
- Le Kip Kip Social Media Campaign: Social media metrics to determine adherence to posting frequency.
Arm/Group | Le Kip Kip Social Media Campaign
Number analyzed (Participants) | NA
Number analyzed (Posts) | 300
Posts
  Content Posting Frequency | 300
  Boosted Post Frequency: number analyzed (Posts) | 119
  Boosted Post Frequency | 100

9. Secondary Outcome: Adoption as Assessed by Number of Views by Unique Users
Description: Service user uptake and engagement with campaign as assessed by number of times each ad was viewed overall and number of video views.
Time Frame: 12 months
Population: As outlined in the protocol, adoption will be assessed using social media metrics and analytics from the number of unique users who have seen the Le Kip Kip Facebook page content at least once.
Measure: Number; unit: views
Units Other Than Participants: Posts
Arm/Group | Le Kip Kip Social Media Campaign
Number analyzed (Participants) | NA
Number analyzed (Posts) | 300
views
  Number of times each ad was viewed | 576384
  Number of times a video was viewed | 44081

10. Secondary Outcome: Adoption as Assessed by Number of Ad Clicks
Description: Service user uptake and engagement with campaign measured via the number of times someone clicked on each ad
Time Frame: 12 months
Population: as for outcome 9
Measure: Number; unit: clicks
Units Other Than Participants: Posts
Arm/Group | Le Kip Kip Social Media Campaign
Number analyzed (Participants) | NA
Number analyzed (Posts) | 300
clicks | 35934

11. Secondary Outcome: Fidelity as Assessed by Programme Logs Completed
Description: Extent to which the social influence campaign was carried out according to plan was measured via trainings, logs of communication with PrEP champions, and community mobilization logs/quality assessments.
Time Frame: 12 months
Population: As outlined in the protocol, the extent to which the social influence campaign was carried out according to plan as assessed via programme logs completed by PrEP champions and community mobilizers.
Measure: Number; unit: percentage of campaign implementers
Units Other Than Participants: Campaign implementers
Arm/Group | Standard of Care | Enhanced Social Media Campaign/PrEP Champions/Community Mobilization
Number analyzed (Participants) | NA | NA
Number analyzed (Campaign implementers) | 0 | 202
percentage of campaign implementers
  Average reporting fidelity among PrEP champions: number analyzed (Campaign implementers) | 0 | 112
  Average reporting fidelity among PrEP champions |  | 49.2
  Average reporting fidelity among community mobilizers: number analyzed (Campaign implementers) | 0 | 90
  Average reporting fidelity among community mobilizers |  | 86.4

ADVERSE EVENTS:
Time Frame: up to 1 year
Arm/Group | Standard of Care | Enhanced Social Media Campaign | Enhanced Social Media Campaign + PrEP Champions | Enhanced Social Media Campaign + Community Mobilization | Enhanced Social Media Campaign + PrEP Champions + Community Mobilization
All-Cause Mortality (participants affected / at risk) | 0/301 | 0/92 | 0/55 | 0/48 | 0/105
Serious Adverse Events (participants affected / at risk) | 0/301 | 0/92 | 0/55 | 0/48 | 0/105
Other Adverse Events (participants affected / at risk) | 0/301 | 0/92 | 0/55 | 0/48 | 0/105

LIMITATIONS AND CAVEATS:
A limitation is using programmatic data to assess PrEP initiation among those accessing HIV testing through TB HIV Care. Since HIV testing and PrEP initiation programmatic data are not linked, we cannot determine the proportion of eligible women who initiate PrEP. Thus, we rely on PrEP initiation counts for the primary outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-20): https://cdn.clinicaltrials.gov/large-docs/20/NCT05417620/Prot_SAP_001.pdf